CLINICAL TRIAL: NCT00797602
Title: A Clinical Outcomes Protocol of Proton Beam Radiation Therapy for Chordomas and/or Chondrosarcomas of the Base of Skull and/or Spine
Brief Title: Proton Therapy for Chordomas and/or Chondrosarcomas
Acronym: CH01
Status: Completed | Type: Observational
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Other Study IDs: UFPTI 0607-CH01
Record Dates: First submitted 2008-11-24; First posted 2008-11-25 (Estimated); Last update posted 2017-08-14 (Actual); Status verified 2017-08

CONDITIONS: Chordomas; Chondrosarcomas
Keywords: Chordomas; Chondrosarcomas; Cancer; Outcomes; Proton radiation
MeSH Terms: conditions — Chordoma; Chondrosarcoma; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Proton Radiation

SUMMARY:
The purpose of this study is to collect information from medical records to see what effects proton beam radiation has on cancer and analyze possible side effects.

DETAILED DESCRIPTION:
Data collection will be obtained from the patient's medical records including initial evaluation, pathology report, dosimetry information, radiotherapy completion records and follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven chordoma or chondrosarcoma.
* Sites: base of skull and/or spine.
* Age 18 years or older.

Exclusion Criteria:

* Previous radiation to the head and neck or brain.
* Evidence of metastatic disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated at a radiation oncology clinic
Sampling Method: Non-Probability Sample
Enrollment: 189 (Actual)
Dates: Start 2007-01; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Collect and analyze outcome data on tumor control. | When each patient has been followed for a minimum of 12 month and then again after 24 months to a maximum of 10 years.

SECONDARY OUTCOMES:
Collect and analyze data on normal tissue morbidity. | When each patient has been followed for a minimum of 12 months and then again after 24 months to a maximum of 10 years.
  Specifically analyzing pituitary, visual and hearing function.

CONTACTS AND LOCATIONS:
Overall Officials: Ronny L Rotondo, MD, Principal Investigator — University of Florida Proton Therapy Institute
Locations (1):
- University of Florida Proton Therapy Institute, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] McMaster ML, Goldstein AM, Bromley CM, Ishibe N, Parry DM. Chordoma: incidence and survival patterns in the United States, 1973-1995. Cancer Causes Control. 2001 Jan;12(1):1-11. doi: 10.1023/a:1008947301735. PMID 11227920
- [Background] Dahlin DC, Unni KK: Bone tumors general aspects and data on 8542 cases, 4th edition. Springfield, IL: Charles C Thomas, 1986, pp 119 - 140.
- [Background] Campbell WM, McDonald TJ, Unni KK, Laws ER Jr. Nasal and paranasal presentations of chordomas. Laryngoscope. 1980 Apr;90(4):612-8. doi: 10.1288/00005537-198004000-00007. PMID 7359980
- [Background] al-Mefty O, Borba LA. Skull base chordomas: a management challenge. J Neurosurg. 1997 Feb;86(2):182-9. doi: 10.3171/jns.1997.86.2.0182. PMID 9010416
- [Background] Pearlman AW, Friedman M. Radical radiation therapy of chordoma. Am J Roentgenol Radium Ther Nucl Med. 1970 Feb;108(2):332-41. No abstract available. PMID 4983924
- [Background] Mendenhall WM, Mendenhall CM, Lewis SB, Villaret DB, Mendenhall NP. Skull base chordoma. Head Neck. 2005 Feb;27(2):159-65. doi: 10.1002/hed.20144. PMID 15641104
- [Background] Fuller DB, Bloom JG. Radiotherapy for chordoma. Int J Radiat Oncol Biol Phys. 1988 Aug;15(2):331-9. doi: 10.1016/s0360-3016(98)90012-8. PMID 2457005
- [Background] Catton C, O'Sullivan B, Bell R, Laperriere N, Cummings B, Fornasier V, Wunder J. Chordoma: long-term follow-up after radical photon irradiation. Radiother Oncol. 1996 Oct;41(1):67-72. doi: 10.1016/s0167-8140(96)91805-8. PMID 8961370
- [Background] Terahara A, Niemierko A, Goitein M, Finkelstein D, Hug E, Liebsch N, O'Farrell D, Lyons S, Munzenrider J. Analysis of the relationship between tumor dose inhomogeneity and local control in patients with skull base chordoma. Int J Radiat Oncol Biol Phys. 1999 Sep 1;45(2):351-8. doi: 10.1016/s0360-3016(99)00146-7. PMID 10487555
- [Background] O'Connell JX, Renard LG, Liebsch NJ, Efird JT, Munzenrider JE, Rosenberg AE. Base of skull chordoma. A correlative study of histologic and clinical features of 62 cases. Cancer. 1994 Oct 15;74(8):2261-7. doi: 10.1002/1097-0142(19941015)74:83.0.co;2-0. PMID 7922977
- [Background] Noel G, Habrand JL, Jauffret E, de Crevoisier R, Dederke S, Mammar H, Haie-Meder C, Pontvert D, Hasboun D, Ferrand R, Boisserie G, Beaudre A, Gaboriaud G, Guedea F, Petriz L, Mazeron JJ. Radiation therapy for chordoma and chondrosarcoma of the skull base and the cervical spine. Prognostic factors and patterns of failure. Strahlenther Onkol. 2003 Apr;179(4):241-8. doi: 10.1007/s00066-003-1065-5. PMID 12707713
- [Background] Berson AM, Castro JR, Petti P, Phillips TL, Gauger GE, Gutin P, Collier JM, Henderson SD, Baken K. Charged particle irradiation of chordoma and chondrosarcoma of the base of skull and cervical spine: the Lawrence Berkeley Laboratory experience. Int J Radiat Oncol Biol Phys. 1988 Sep;15(3):559-65. doi: 10.1016/0360-3016(88)90295-7. PMID 3138208
- [Background] Hug EB, Sweeney RA, Nurre PM, Holloway KC, Slater JD, Munzenrider JE. Proton radiotherapy in management of pediatric base of skull tumors. Int J Radiat Oncol Biol Phys. 2002 Mar 15;52(4):1017-24. doi: 10.1016/s0360-3016(01)02725-0. PMID 11958897
- [Background] Austin JP, Urie MM, Cardenosa G, Munzenrider JE. Probable causes of recurrence in patients with chordoma and chondrosarcoma of the base of skull and cervical spine. Int J Radiat Oncol Biol Phys. 1993 Feb 15;25(3):439-44. doi: 10.1016/0360-3016(93)90065-4. PMID 8436522
- [Background] Fagundes MA, Hug EB, Liebsch NJ, Daly W, Efird J, Munzenrider JE. Radiation therapy for chordomas of the base of skull and cervical spine: patterns of failure and outcome after relapse. Int J Radiat Oncol Biol Phys. 1995 Oct 15;33(3):579-84. doi: 10.1016/0360-3016(95)02014-3. PMID 7558946
- [Background] Parsons JT, Bova FJ, Fitzgerald CR, Mendenhall WM, Million RR. Radiation optic neuropathy after megavoltage external-beam irradiation: analysis of time-dose factors. Int J Radiat Oncol Biol Phys. 1994 Nov 15;30(4):755-63. doi: 10.1016/0360-3016(94)90346-8. PMID 7960976
- [Background] Parsons JT, Bova FJ, Fitzgerald CR, Mendenhall WM, Million RR. Radiation retinopathy after external-beam irradiation: analysis of time-dose factors. Int J Radiat Oncol Biol Phys. 1994 Nov 15;30(4):765-73. doi: 10.1016/0360-3016(94)90347-6. PMID 7960977
- [Background] Bhandare N, Monroe AT, Morris CG, Bhatti MT, Mendenhall WM. Does altered fractionation influence the risk of radiation-induced optic neuropathy? Int J Radiat Oncol Biol Phys. 2005 Jul 15;62(4):1070-7. doi: 10.1016/j.ijrobp.2004.12.009. PMID 15990010